CLINICAL TRIAL: NCT00126477
Title: The Quality of Life of Adult Survivors Who Received a Marrow Transplant as a Child
Brief Title: Quality of Life of Adult Cancer Survivors Who Have Undergone a Previous Bone Marrow or Peripheral Stem Cell Transplant for a Childhood Hematologic Cancer
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 1098.00; FHCRC-1098.00; CDR0000434793 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Quality of Life
Keywords: quality of life; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; juvenile myelomonocytic leukemia; childhood Hodgkin lymphoma; childhood lymphoblastic lymphoma; childhood large cell lymphoma; childhood small noncleaved cell lymphoma; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma | interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: cognitive assessment
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Studying quality of life in cancer survivors may help determine the long-term effects of hematologic cancer and may help improve the quality of life for future cancer survivors.

PURPOSE: This clinical trial is studying the quality of life of adult cancer survivors who have undergone a previous bone marrow or peripheral stem cell transplant for a childhood hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the extent to which adult cancer survivors who have undergone prior bone marrow or peripheral blood stem cell transplantation for a pediatric hematologic malignancy require ongoing health care and whether these needs change with increasing time after transplantation.
* Correlate physical capabilities, body image, physical limitations, including sexuality issues which alter or influence lifestyle, with time after transplantation in these patients.
* Determine whether cognitive abilities relative to memory and neurobehavioral ratings change with increasing time after transplantation in these patients.
* Correlate social and relationship abilities with length of time after transplantation in these patients.

OUTLINE: Patients and siblings complete a self-report quality of life questionnaire, including outcome assessments of neuroendocrine function, cognitive abilities, physical capability, and psychosocial behavior.

PROJECTED ACCRUAL: Approximately 750 patients (375 adult cancer survivors [case group] and 375 siblings [control group]) will be accrued for this study within 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Case group

  * Previously treated with an allogeneic, unrelated, syngeneic, or autologous bone marrow or peripheral blood stem cell transplantation for a hematologic malignancy ≥ 5 years ago while enrolled on 1 of the following protocols:

    * FHCRC-160.06
    * FHCRC-179.07T
    * FHCRC-446.03T
    * FHCRC-661.04
    * FHCRC-697.00
    * FHCRC-796.00
    * FHCRC-843.00
  * Disease-free survivor
  * Under 18 years of age at time of transplantation
  * Any prior preparative regimen allowed
* Control group

  * Sex-matched sibling within 5 years of patient's age*
  * No chronic illnesses (e.g., cancer, diabetes, or asthma) that require medication
  * No allergies that limit physical activity NOTE: *If such a sibling is not available, but another sibling is available, then that sibling would be asked to nominate a friend or relative of the same gender as the patient who is also within 5 years of the patient's age; the patient must consent in order for the control subject to participate

PATIENT CHARACTERISTICS:

Age

* See Disease Characteristics
* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Must be able to speak, read, and write English

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 1996-03; Primary Completion 2007-04 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Neuroendocrine status of disease-free childhood transplant patients at 5 years after transplant and ≥ age 18
Cognitive capability of disease-free childhood transplant patients at 5 years after transplant and ≥ age 18
Physical capability of disease-free childhood transplant patients at 5 years after transplant and ≥ age 18
Psychosocial status of disease-free childhood transplant patients at 5 years after transplant and ≥ age 18

CONTACTS AND LOCATIONS:
Overall Officials: Jean E. Sanders, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States